CLINICAL TRIAL: NCT05084690
Title: Mirror Illusion Training to Improve Contralateral Arm Strength
Brief Title: Mirror Illusion Training and Cross-education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Joshua Carr, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-102
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Exercise Therapy; Weight Lifting
Keywords: Strength training; Mirror visual feedback

STUDY DESIGN:
Intervention Model Description: Randomized, two arm parallel experimental and control groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training control group (Active Comparator): The resistance training control group will perform unilateral resistance training on their dominant arm. The training will be performed twice per week for four weeks totaling eight training sessions.
  Interventions: Other: Unilateral resistance training
- Resistance training with mirror illusion group (Experimental): The resistance training with mirror illusion group will perform unilateral resistance training on their dominant arm. During training, they will view a mirror illusion of their exercising arm over their opposite, non-exercising arm. The training will be performed twice per week for four weeks totaling eight training sessions.
  Interventions: Other: Unilateral resistance training; Other: Illusionary mirror visual feedback

INTERVENTIONS:
Other: Unilateral resistance training — Unilateral resistance training of the elbow flexors
Other: Illusionary mirror visual feedback — Modified Ramachandran's mirror box
  Arms: Resistance training with mirror illusion group

SUMMARY:
Cross-education describes the transfer of motor performance to the opposite limb following unilateral training and is primarily explained by adaptations within the brain. The mirror training hypothesis suggests that illusionary mirror visual feedback may augment the cross-education of strength to the untrained, contralateral limb. The purpose of this project is to examine how the use of illusionary mirror visual feedback shapes the neuromuscular adaptations that occur for both limbs during unilateral (single-limb) strength training. Our hypothesis is that mirror training will augment the level of cross-education for the untrained arm.

DETAILED DESCRIPTION:
Recent empirical evidence shows a heightened level of strength transfer with the use of illusionary mirror visual feedback, but this was shown for the small muscles of the wrist during isokinetic training. It is unknown if larger, multi-joint muscles respond favorably to mirror training in practical settings. A randomized controlled study design will allocate approximately 20 participants into two groups. One group will perform unilateral strength training with illusionary mirror visual feedback (Mirror) and the other will perform the same unilateral strength training but without a mirror (No-Mirror). The intervention will involve four weeks of unilateral strength training performed twice weekly at high intensities (>80%1RM).

ELIGIBILITY:
Inclusion Criteria:

* right-hand dominance
* no previous strength training of upper body last 3 months
* no injuries or recent surgeries of the upper limbs
* willingness to adhere to the strength training requirements of the study

Exclusion Criteria:

* current use of hormone replacement therapy
* pregnancy/breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-08-19 (Estimated); Study Completion 2023-08-19 (Estimated)

PRIMARY OUTCOMES:
Change in dynamic muscle strength for the trained and untrained arm | Baseline (week 0) post-training (week 5)
  Dynamic 1-repetition maximum (lbs)
Change in isometric muscle strength for the trained and untrained arm | Baseline (week 0) post-training (week 5)
  Isometric maximal voluntary contraction
Change in lean mass for the trained and untrained arm | Baseline (week 0), mid-training (week 2), post-training (week 5)
  DEXA (g)
Change in muscle thickness for the trained and untrained arm | Baseline (week 0), mid-training (week 2), post-training (week 5)
  Ultrasound muscle thickness (cm)
Change in muscle activation for the trained and untrained arm | Baseline (week 0) post-training (week 5)
  Electromyographic amplitude (volts)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Carr, Principal Investigator — Texas Christian University
Locations (2):
- United States (2):
  - TCU Neuromuscular Physiology Laboratory, Fort Worth, Texas
  - TCU RIC, Fort Worth, Texas